CLINICAL TRIAL: NCT03664154
Title: Stress and Feeding (SAFE): A Pilot Intervention for Mothers and Their Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HM20013532
Record Dates: First submitted 2018-08-24; First posted 2018-09-10 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Feeding Behavior; Preterm Infant; Stress; Mother-Infant Interaction
MeSH Terms: conditions — Feeding Behavior; Premature Birth

STUDY DESIGN:
Intervention Model Description: A one-group longitudinal repeated measures design. Data will be collected at baseline, 8-weeks, 12-weeks, and 16-weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stress and Feeding (SAFE) (Experimental): The SAFE intervention is grounded in a general theory of guided participation (GP) that posits learning will be facilitated by an emotionally regulated state of the mother. Efforts to help mothers manage stress will better position them to learn and attend to feeding their infants. GP links the two components: stress management (SM) and guided feeding (GF). SM provides skills to manage perceived stress and regulate emotion. GF provides education with skill building to help mothers become more sensitive and responsive to their infant. SAFE is delivered through a secure, password-protected responsive website with practice opportunities.
  Interventions: Behavioral: Stress and Feeding (SAFE)

INTERVENTIONS:
Behavioral: Stress and Feeding (SAFE) — The Stress Management component of the intervention acknowledges the mind-body connection between stress and adverse outcomes and consists of four web-based modules based on Lazarus and Folkman's Transactional Model of Stress and Coping designed to improve health outcomes.
  The Guided Feeding component of the intervention is based on the synactive theory of development. The synactive theory of development provides insight in to reading the physiological and behavioral cues of infants born preterm and involves weekly viewing of video clips of adaptive and maladaptive feeding behaviors of mothers and infants, practice opportunities, and follow-up phone calls.

SUMMARY:
A majority of mothers experience high stress levels and associated symptoms of anxiety, depressive symptoms, and sleep disruption during the NICU hospitalization and continuing after hospital discharge. Given preterm infant feeding is one of the most stressful things the new mother will face and given the harmful nature of stress on maternal and infant health, it is important an intervention focuses on both of these concerns: infant feeding and maternal stress. Therefore, the purpose of this research study is two-fold. First, the investigators will examine how practical and acceptable it is for mothers of preterm infants to participate in Stress And FEeding (SAFE) intervention and collect biological stress measures from mothers and their preterm infant's saliva (spit). The intervention is designed to reduce stress and improve maternal feeding interaction. The second purpose of this study is to examine changes before and after using the intervention on mother and infant outcomes over 16-weeks.

DETAILED DESCRIPTION:
Descriptive statistics will be computed for demographic and outcome variables. The number of mother/infant dyads recruited but not enrolled will be tracked. If provided, reasons for non-participation will be noted. Enrolled dyads will be tracked and monitored for the number of times the interventions are used and completeness of study data. Acceptability and burden will be assessed by theme analysis of the responses to the interview by the mPI's using traditional strategies of reading and re-reading the transcripts, coding participant responses using their language, and developing categories and subcategories to create a structure for considering acceptability will be completed.. Finally, perceptions of usefulness and satisfaction of the mothers will be assessed by looking at frequencies of Likert responses.

Means and standard errors of the maternal stress and feeding behavior variables will be estimated and graphed across the data collection time points. Although the sample size is small, it is anticipated the mixed effects linear model will be used to assess and quantify changes across time. This model will include a random effect for participant and a fixed effect for time. The model is flexible enough to model potential cofactors, such as age at birth. The study will track the number of successfully obtained, transported, processed and stored samples and compare those number to the proposed maternal and infant cortisol collections.

ELIGIBILITY:
Maternal Inclusion Criteria:

* English-speaking and reading
* Given birth to preterm infant < 35-weeks gestation
* Has access to internet
* Lives within 50-mile radius of hospital

Infant Inclusion Criteria:

* Born less than 35 week gestation
* No congenital anomalies that could interfere with feeding (e.g., diaphragmatic hernia, cleft lip/palate tracheoesophageal fistula, and cardiac anomalies

Maternal Exclusion Criteria:

* Chronic neuroendocrine or immunologic condition
* Currently using guided imagery or other mind-body techniques such as meditation
* Psychiatric disorder involving a history of dissociative disorders, borderline personalities, and psychotic pathology

Infant Exclusion Criteria:

* Grade III or IV intraventricular hemorrhage
* Surgical necrotizing enterocolitis

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women who have given birth to a premature infant (either male or female)
Enrollment: 10 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Ease of recruitment of participants | 12-months after study opens to enrollment
  Number of mother-infant dyads recruited, with a goal of 15
Track non-participation | 16-weeks after start of intervention
  Track reasons for non-participation via self-report
Adherence | 16-weeks after start of intervention
  Adherence will be assessed by tracking the number of times the interventions are used
Data collection completeness | 16-weeks after start of intervention
  Percent of participants with complete data collection at end of study, with a goal of >75% of patients
Appraisal of SAFE's degree of inconvenience | 16-weeks after start of intervention
  The participants appraisal of inconvenience will be measured through a semi-structured interview and will be described qualitatively
Satisfaction with intervention | 16-weeks after start of intervention
  The participants satisfaction with the intervention will be measured using a 26-item Likert scale where 1 represents being not at all satisfied to 5 being very much satisfied.

SECONDARY OUTCOMES:
Change in maternal stress | Baseline to 16-weeks post-baseline
  Paper and pencil questions asking about degree to which situations in an individual's life are appraised as stressful and asking about common problems mothers with young children face daily, with higher scores indicating more stress
Changes in mother biological stress | Baseline to 16-weeks post-baseline
  Biological stress will be assessed by changes in salivary cortisol of mother (an indicator of mother and infant stress)
Changes in infant biological stress | Baseline to 16-weeks post-baseline
  Biological stress will be assessed by changes in salivary cortisol of infant (an indicator of mother and infant stress)
Changes in mother-infant feeding behaviors | Baseline to 16-weeks post-baseline
  Mother and infant feeding behaviors will be assessed using the Parent-Child Early Relational Assessment (PCERA). The PCERA is scored on a 5-point Likert scale on quality, intensity, or amount, and duration of behavior where 1 represents negative behavior of clinical concern and 5 represents regulated, adaptive behavior

OTHER OUTCOMES:
Practicability of collecting cortisol | 16-weeks after start of intervention
  Practicability will be assessed by tracking the number of successfully obtained, transported, processed, and stored cortisol samples

CONTACTS AND LOCATIONS:
Overall Officials: Lisa F Brown, PhD, RN, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers.

REFERENCES:
- [Background] Als, H. (1986). A synactive model of neonatal behavioral organization: framework for the assessment of neurobehavioral development in the premature infant and for support of infants and parents in the neonatal intensive care environment. Physical & Occupational Therapy in Pediatrics, 6(2-3), 3-53. http://doi.org/10.1080/J006v06n03_02
- [Background] Als H, Gilkerson L. The role of relationship-based developmentally supportive newborn intensive care in strengthening outcome of preterm infants. Semin Perinatol. 1997 Jun;21(3):178-89. doi: 10.1016/s0146-0005(97)80062-6. PMID 9205974
- [Background] Lazarus, R. S., & Folkman, S. (1984). Stress, Appraisal, and Coping. New York, NY: Springer Publishing.
- [Background] Pridham KF. Guided participation and development of care-giving competencies for families of low birth-weight infants. J Adv Nurs. 1998 Nov;28(5):948-58. doi: 10.1046/j.1365-2648.1998.00814.x. PMID 9840866
- [Background] Pridham K, Brown R, Clark R, Limbo RK, Schroeder M, Henriques J, Bohne E. Effect of guided participation on feeding competencies of mothers and their premature infants. Res Nurs Health. 2005 Jun;28(3):252-67. doi: 10.1002/nur.20073. PMID 15884024
- [Background] Jung JW. Apprenticeship in thinking: cognitive development in social context (barbara rogoff). Korean J Med Educ. 2009 Jun;21(2):197-8. doi: 10.3946/kjme.2009.21.2.197. Epub 2009 Jun 30. No abstract available. PMID 25813118
- [Background] Rogoff, B. (2003). The cultural nature of human development. New York: Oxford University Press.
- [Background] Schroeder M, Pridham K. Development of relationship competencies through guided participation for mothers of preterm infants. J Obstet Gynecol Neonatal Nurs. 2006 May-Jun;35(3):358-68. doi: 10.1111/j.1552-6909.2006.00049.x. PMID 16700685
- [Background] Wethington, E., Glanz, K., & Schwartz, M. (2015). Stress, coping and health behavior. In K. Glanz, B. K. Rimer, & K. Viswanath (Eds.), Health Behavior: theory, Research & Practice (5th ed., pp. 223-242). San Francisco, CA: Jossey-Bass.
- [Background] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405

DOCUMENTS (1):
  • Informed Consent Form (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT03664154/ICF_000.pdf